CLINICAL TRIAL: NCT04715737
Title: The Differential Effects of Intranasal Vasopressin and Oxytocin on Attention Control
Brief Title: Differential Effects of Vasopressin and Oxytocin on Attention Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-76
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Vasopressin; Oxytocin; Eye-tracking; Attention control
MeSH Terms: conditions — Diabetes Insipidus | interventions — Vasopressins; Oxytocin

STUDY DESIGN:
Intervention Model Description: Between-subject randomized placebo-controlled double-blind pharmacological eye-tracking design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vasopressin (Experimental): Vasopressin (20IU) intranasally
  Interventions: Drug: Vasopressin
- Oxytocin (Experimental): Oxytocin (24IU) intranasally
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo intranasally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vasopressin — Administration of vasopressin (20IU) intranasally
  Arms: Vasopressin
Drug: Oxytocin — Administration of oxytocin (24IU) intranasally
  Arms: Oxytocin
Drug: Placebo — Administration of placebo intranasally
  Arms: Placebo

SUMMARY:
The main aim of the present study is to investigate whether intranasal vasopressin (20IU) and oxytocin (24IU) have differential effects on attention control in a social-emotional saccade/antisaccade eye-tracking paradigm.

DETAILED DESCRIPTION:
Previous studies have demonstrated intranasal vasopressin and oxytocin's divergent effects on social behavior and emotion processing such as empathy and negative emotion processing, however, it remains unclear whether vasopressin and oxytocin treatment would have differential effects on attention processing to social stimuli. Based on the previous registered studies (ClinicalTrials.gov ID: NCT04493554 and NCT03486925) from our group using a validated emotional anti-saccade task with social stimuli (emotional faces) and non-social stimuli (oval shape) have separately explored intranasal vasopressin and oxytocin's modulatory effects on attention processing, the present study aims to conduct a secondary analysis of the previously acquired data to directly compare vasopressin and oxytocin's effects on attention control to social emotional stimuli. To this end data from subjects who underwent intranasal oxytocin administration (n = 33; NCT03486925) will be compared with data from subjects who underwent intranasal vasopressin or placebo administration (n = 39, or 45 respectively; NCT04493554). To further control for non-treatment related factors the intranasal placebo groups from the previous studies (ClinicalTrials.gov ID: NCT04493554 and NCT03486925) will be compared with respect to primary and secondary outcome measures of the trial, in particular general and emotion-specific effects on attentional control.

ELIGIBILITY:
Inclusion Criteria:

* Male, healthy participants
* Non smokers

Exclusion Criteria:

* Previous or current medical, psychiatric, neurological disorder
* Regular medication
* Use of any psychoactive substances in the 24 hours before experiment

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Differential effects of intranasal vasopressin and oxytocin administration on saccade/antisaccade latencies towards social (facial) versus non-social (shape) stimuli | Time Frame: 45 minutes - 100 minutes after treatment
  Comparison between social-specific saccade/antisaccade latencies (in milliseconds) between the vasopressin, oxytocin and placebo treatment conditions
Differential effects of intranasal vasopressin and oxytocin administration on error rates of saccade/antisaccade for social (facial) versus non-social (shape) stimuli | Time Frame: 45 minutes - 100 minutes after treatment
  Comparison between social-specific error rates of saccade/antisaccade between the vasopressin, oxytocin and placebo treatment conditions

SECONDARY OUTCOMES:
Emotion-specific effects of vasopressin and oxytocin administration on saccade/antisaccade latencies towards the separate facial emotions | Time Frame: 45 minutes - 100 minutes after treatment
  Comparison between emotion-specific saccade/antisaccade latencies (in milliseconds) between the vasopressin, oxytocin and placebo treatment conditions
Emotion-specific effects of vasopressin and oxytocin administration on saccade/antisaccade error rates for the separate facial emotions | Time Frame: 45 minutes - 100 minutes after treatment
  Comparison between emotion-specific saccade/antisaccade error rates between the vasopressin, oxytocin and placebo treatment conditions

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China (UESTC)
Locations (1):
- University of Electronic Science and Technology of China (UESTC), Sichuan, Chengdu, China

IPD SHARING:
Plan to Share IPD: No